CLINICAL TRIAL: NCT00896519
Title: An Open Label, Multicenter, Non Randomized Phase II Study to Evaluate Antitumor Efficacy and Safety of GM-CSF (Sargramostim, Leukine®) Associated With RCHOP Chemotherapy and Rituximab (MabThera®) Maintenance in Patients With First-line Advanced Follicular Non Hodgkin's Lymphoma
Brief Title: GM-CSF, Rituximab, and Combination Chemotherapy in Treating Patients With Previously Untreated Advanced Follicular Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: French Innovative Leukemia Organisation (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: GOELAMS-FL2008-RCHOP-GM; CDR0000637105 (Registry Identifier: PDQ (Physician Data Query)); FL2008-RCHOP-GM; EUDRACT2007-007056-33; RECF0907
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2009-07

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; sargramostim; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Gene Expression Profiling; Gene Rearrangement; Polymerase Chain Reaction

INTERVENTIONS:
Biological: rituximab
Biological: sargramostim
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Genetic: gene expression analysis
Genetic: gene rearrangement analysis
Genetic: polymerase chain reaction
Other: R-CHOP regimen
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as GM-CSF, may cause the body to make more blood cells and help it recover from the side effects of rituximab and combination chemotherapy.

PURPOSE: This phase II trial is studying how well giving GM-CSF together with rituximab and combination chemotherapy works in treating patients with previously untreated advanced follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the overall objective tumor response rate (complete and partial response rates) in patients with previously untreated advanced follicular non-Hodgkin lymphoma treated with sargramostim (GM-CSF) and R-CHOP.

Secondary

* To evaluate the time to progression.
* To evaluate the overall survival.
* To evaluate the duration of response.
* To evaluate the time to next treatment.
* To evaluate the safety profile of GM-CSF in combination with R-CHOP.
* To evaluate the influence of FcγR polymorphisms on clinical response.
* To monitor FcγR expressing cells in peripheral blood during treatment.
* To monitor the molecular biological marker bcl-2 [t(14;18)] in peripheral blood and bone marrow by quantitative PCR assay.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive R-CHOP comprising rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1 and oral prednisone on days 1-5. Patients also receive sargramostim (GM-CSF) subcutaneously (SC) on days 2-6. Treatment repeats every 21 days for up to 6 courses. Patients then receive rituximab IV on day 1 and GM-CSF SC on days 1-5. Treatment with rituximab and GM-CSF repeats every 21 days for 2 courses. Patients achieving complete or partial response proceed to maintenance therapy.
* Maintenance therapy: Patients receive rituximab IV on day 1 and GM-CSF SC on days 1-5. Treatment repeats every 2 months for 12 courses.

Blood and bone marrow samples are collected at baseline and periodically during study for analysis of FcγR expression by immunophenotyping and bcl-2 rearrangement by quantitative PCR.

After completion of study therapy, patients are followed every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular non-Hodgkin lymphoma

  * Grade 1-3a disease
  * Advanced disease
* Has undergone initial lymph node biopsy within the past 4 months
* At least 1 measurable lesion
* Bulky disease, as defined by the following GELF criteria:

  * Nodal or extranodal mass > 7 cm in its greatest diameter
  * Involvement of ≥ 3 nodal sites (each with a diameter > 3 cm)
  * B symptoms
  * Elevated serum LDH or β2-microglobulin
  * Splenic enlargement
  * Compression syndrome
  * Pleural and/or peritoneal effusion
* No transformation to high-grade follicular lymphoma (secondary to low-grade follicular lymphoma)
* No prior or concurrent CNS disease (i.e., CNS lymphoma or lymphomatous meningitis) NOTE: A new classification scheme for adult non-Hodgkin lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* ANC ≥ 1,000/mm^3*
* Platelet count ≥ 100,000/mm^3*
* Hemoglobin ≥ 8.0 g/dL*
* Total bilirubin ≤ 2.0 mg/dL*
* AST ≤ 3 times upper limit of normal*
* Serum creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* No known HIV infection
* No active hepatitis B or C infection
* No serious underlying medical condition that would preclude study participation (e.g., ongoing infection, uncontrolled diabetes mellitus, gastric ulcer, active autoimmune disease, or heart failure)
* No known sensitivity or allergy to murine products
* No other prior or concurrent malignancies except nonmelanoma skin cancer or adequately treated in situ cervical cancer
* No other co-existing medical or psychological condition that would preclude study participation or ability to give informed consent NOTE: *Unless abnormalities are related to lymphoma

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior treatment for follicular lymphoma, including steroids or radiotherapy
* More than 4 weeks since prior corticosteroids unless administered at a dose equivalent to < 20 mg/day of prednisone
* More than 28 days since prior major surgery (excluding lymph node biopsy)
* More than 30 days since prior treatment in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Overall objective tumor response rate

SECONDARY OUTCOMES:
Time to treatment progression
Overall survival
Duration of response
Time to next treatment
Safety profile
Influence of FcγR polymorphisms on clinical response and overall survival
Monitoring of FcγR expressing cells during treatment
Quantitative monitoring of the molecular biological marker bcl-2 in peripheral blood and bone marrow by PCR assay

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rossi, MD, PhD, Principal Investigator — Hopital Lapeyronie-CHU Montpellier